



## **Participant Consent Form**

Study Title: Art therapy to address hospital clinician burnout and psychosocial distress: a randomised controlled trial (CHArt) IRAS: 316097 Participant identification number for this trial: Name of Researcher: Megan Tjasink Please initial boxes 1. I have read the Information Sheet: Version 1.2: 24.10.2023 for the above study. I have been emailed or given a hard copy of the document to keep. 2. I have had the opportunity to consider the information and ask questions about the above study. I am satisfied with the responses I received to questions I asked. 3. I understand that my participation is voluntary and that I am free to withdraw from the study at any time, without having to give a reason, and without my legal rights being affected. 4. I understand that participation in this research involves completing questionnaires and that direct quotations may be reproduced in reports and publications, but all identifying information will be removed. 5. I understand that relevant sections of data collected during the study may be looked at by individuals from Queen Mary University of London, from regulatory authorities or from Barts Health NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to these records. 6. I understand that participation involves my artwork (made during the workshops) being photographed, and that these may be reproduced in reports and publications, but all identifying information will be removed. 7. I agree to being contacted with the option to take part in future related research after the end of the study. 8. I agree to take part in the above study. Name of Participant Signature Date Name of Person taking consent Date Signature